CLINICAL TRIAL: NCT01393262
Title: Orthopaedic Hand Service Data Repository
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Neal Chung-Jen Chen, Principal Investigator; Director of Research, Hand Service, Massachusetts General Hospital
Other Study IDs: 2009-P-001019
Record Dates: First submitted 2011-07-11; First posted 2011-07-13 (Estimated); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Non-traumatic and Traumatic Health Issues

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Healthy Escort
- Hand Service patient

SUMMARY:
The purpose of the research is to investigate multiple facets of non-traumatic and traumatic health issues. The majority of our research deals with mind-body aspects of health. The investigators often correlate different psychological measures against one another or match psychological and depression scores against standard of care objective measurements (grip strength and range of motion).

The data repository also serves to streamline our studies and amalgamate many studies that are no more than minimal risk and do not involve randomization in any way.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years
* Patients presenting to Hand Service for traumatic or non-traumatic issues.
* English Speaking

Exclusion Criteria:

* under 18 years
* vulnerable population

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All individuals will be over the age of 18 and English speaking, excluding vulnerable populations (mental disabilities, prisoners etc.). Patients may be traumatic or non-traumatic.
Sampling Method: Probability Sample
Enrollment: 9620 (Actual)
Dates: Start 2009-11 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neal Chen, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States